CLINICAL TRIAL: NCT06621017
Title: A Randomized, Placebo-Controlled, Double-Blind, Parallel-Group Study Evaluating the Efficacy, Safety, and Pharmacokinetics of Daily Administrations of the GLP-1 Analogue ROSE-010 on Appetite and Food Intake in Overweight and Obese Subjects
Brief Title: Effect of GLP-1 Analogue ROSE-010 on Appetite in Overweight and Obese Subjects
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Rose Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RP-24-02
Record Dates: First submitted 2024-09-26; First posted 2024-10-01 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Obesity; Overweight
Keywords: GLP-1; ROSE-010; Obesity; Overweight; Appetite depressant; Pharmacokinetics
MeSH Terms: conditions — Obesity; Overweight; Anorexia | interventions — glucagon-like peptide (7-37), valyl(10)-

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Placebo (Placebo Comparator): Saline solution
  Interventions: Drug: Placebo
- ROSE-010 99 mcg (Experimental): ROSE-010 solution, 99 mcg, 0.5 ml
  Interventions: Drug: ROSE-010 99 mcg
- ROSE-010 150 mcg (Experimental): ROSE-010 solution, 150 mcg, 0.5 ml
  Interventions: Drug: ROSE-010 150 mcg

INTERVENTIONS:
Drug: ROSE-010 99 mcg — Sub-cutaneous injection of ROSE-010 solution
  Arms: ROSE-010 99 mcg
Drug: Placebo — Sub-cutaneous injection of saline solution
  Arms: Placebo
Drug: ROSE-010 150 mcg — Sub-cutaneous injection of ROSE-010 solution
  Arms: ROSE-010 150 mcg

SUMMARY:
The primary objective of this study is to assess the efficacy of ROSE-010 on food intake in female subjects with overweight and obesity.

The secondary objectives of this study are the following:

* To assess the efficacy of ROSE-010 on hunger;
* To assess the efficacy of ROSE-010 on satiety;
* To assess the efficacy of ROSE-010 on prospective consumption;
* To assess the efficacy of ROSE-010 on desire to eat;
* To assess the efficacy of ROSE-010 on palatability;
* To characterize the pharmacokinetics (PK) of ROSE-010 following subcutaneous (SC) administration on Day 1 and Day 7; and
* To evaluate safety and tolerability of SC administrations of ROSE-010 to overweight and obese subjects.

DETAILED DESCRIPTION:
This is a randomized, placebo-controlled, double-blind, parallel-group Phase 2 study evaluating the efficacy, safety, and PK of daily administrations of the GLP-1 analogue ROSE-010 on appetite and food intake in overweight and obese female subjects. The study is planned to include 3 parallel groups, as follows:

Group 1: 99 mcg ROSE-010 (15 subjects) administered SC once daily for 7 consecutive days.

Group 2: 150 mcg ROSE-010 (15 subjects) administered SC once daily for 7 consecutive days.

Group 3: Placebo (10 subjects) administered SC once daily for 7 consecutive days.

On Day 1, subjects will be randomized to receive ROSE-010 or placebo. Study drug will be administered SC once daily (30 minutes before lunch) for 7 consecutive days (Days 1 to 7). Assessments of hunger, satiety, prospective consumption, desire to eat, palatability, and nausea will be performed. Blood samples will be collected to evaluate PK.

ELIGIBILITY:
Inclusion Criteria:

1. Body mass index greater or equal to 27 and less than nor equal to 35 kg/m2 at Screening.
2. Good health, as assessed by the Investigator, based on medical, surgical, and psychiatric history, physical examination, 12-lead electrocardiogram (ECG), vital sign assessments, and clinical laboratory evaluations at Screening and Check-In.
3. Subjects must have a negative serum pregnancy test result at Screening and at Check-In and must not be pregnant, lactating, or planning a pregnancy from the Screening Visit to 30 days after the last dose of study drug.
4. Female subjects of non-childbearing potential must be either surgically sterile (ie, had a hysterectomy, bilateral tubal ligation, bilateral salpingectomy, and/or bilateral oophorectomy at least 26 weeks prior to Screening) or postmenopausal (ie, have experienced spontaneous amenorrhea for at least 2 years, with a follicle-stimulating hormone level in the postmenopausal range at Screening based on the central laboratory's ranges).
5. Subjects of childbearing potential (ie, ovulating, premenopausal, and not permanently surgically sterile) with male partners will be included if they are either sexually inactive (complete abstinence from heterosexual activity if in line with the subject's preferred and usual lifestyle) for at least 30 days prior to the first dose of study drug and agree to continue complete abstinence for at least 30 days after the last administration of study drug, or, if sexually active, agree to use a medically accepted contraceptive regimen during their participation in the study and for at least 30 days after the last administration of study drug.

Exclusion Criteria:

1. Clinically significant or active gastric emptying abnormality (eg, gastroparesis or gastric outlet obstruction, intestinal obstruction, or any gastrointestinal [GI] motility disorders); malabsorption, including chronic constipation/diarrhea, celiac disease, inflammatory bowel disease, or bowel resection; or chronic use of drugs that directly affect GI motility (eg, anticholinergics, 5-hydroxytryptamine [serotonin] antagonists, opiates).
2. Obesity induced by other endocrinologic disorders (eg, Cushing syndrome, acromegaly, inadequately treated hypothyroidism) or diagnosed monogenic or syndromic forms of obesity (eg, melanocortin 4 receptor deficiency or Prader-Willi syndrome).
3. Thyroid disease that is not controlled (thyroid-stimulating hormone outside normal range at Screening).
4. Symptomatic gallbladder disease within the past 2 years or history of cholecystectomy.
5. History or presence of chronic pancreatitis or presence of acute pancreatitis within 6 months before Screening.
6. A history of Major Depressive Disorder within the last 2 years.
7. Any lifetime history of a suicide attempt.
8. Previous bariatric surgery, procedure for obesity, or GI surgery altering GI passage, motility, and/or nutrient absorption or recent (within 6 months of Screening) changes in body weight (greater or equal to 5%) due to dieting, including commercial weight loss programs, or pharmacologic treatment.
9. Currently on or planning to participate in any weight loss regimen during the course of the study.
10. Personal or family history of medullary thyroid carcinoma or multiple endocrine neoplasia type 2.
11. History of malignancy, except the following: curatively resected basal cell or squamous cell skin cancers, cervical cancer in situ, or resected colorectal polyps more than 5 years prior to Screening.
12. Abnormal fasting blood glucose (ie, greater than 125 mg/dL) at Screening or Check-In and/or HbA1c (greater than 6.4%) at Screening, or prior history/diagnosis of any type of diabetes mellitus (eg, type 1, type 2, or gestational).
13. Use of any prescribed or over-the-counter (OTC) medication other than approved contraceptives within 14 days or 5 half-lives (whichever is longer) prior to dosing on Day 1 and throughout the study.

    Note: Following study drug administration, medications used for the treatment of adverse events (AEs) may be allowed at the discretion of the Investigator or designee.
14. Any glucagon-like peptide-1 (GLP-1) receptor agonist, GLP-1/glucose-dependent insulinotropic polypeptide dual agonist (eg, tirzepatide), or any prescription or OTC medications intended for weight loss or with a potential impact on weight and appetite regulation (eg, stimulant medications) within 6 months of Screening.
15. Known allergy to any ingredient of ROSE-010 or any history of severe allergic reaction (including drugs, food, insect bites, or environmental allergens).

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2024-09-26 (Actual); Primary Completion 2025-02-27 (Actual); Study Completion 2025-02-27 (Actual)

PRIMARY OUTCOMES:
Food consumption | 30 minutes
  The amount of food (weight and energy content) consumed during lunch after administration of ROSE-010 at 2 dose levels compared to placebo.

SECONDARY OUTCOMES:
Hunger | 6.5 hours
  Hunger score on a visual analogue scale (VAS) (0 to 100 mm)
Satiety | 6.5 hours
  Satiety score on a VAS (0 to 100 mm)
Prospective consumption | 6.5 hours
  Prospective consumption score on a VAS (0 to 100 mm)
Desire to eat | 6.5 hours
  Desire to eat score on a VAS (0 to 100 mm)
Palatability | 30 minutes
  Palatability (tastiness) score on a VAS (0 to 100 mm)
Nausea | 6.5 hours
  Incidence and severity of nausea on a VAS (0 to 100 mm)
Plasma PK analysis of ROSE-010 Elimination | 7 days
  Plasma PK analysis of ROSE-010: Terminal phase elimination half-life.
Plasma PK analysis of ROSE-010 Cmax | 7 days
  Plasma PK analysis of ROSE-010: maximum serum concentration (Cmax).
Plasma PK analysis of ROSE-010 Cmax Time | 7 days
  Plasma PK analysis of ROSE-010: Time to Cmax.
Plasma PK analysis of ROSE-010 Concentration over time | 7 days
  Plasma PK analysis of ROSE-010: Area under the plasma concentration-time curve.

CONTACTS AND LOCATIONS:
Locations (1):
- Medpace Clinical Pharmacology, Cincinnati, Ohio, United States

IPD SHARING:
Plan to Share IPD: No